CLINICAL TRIAL: NCT05715931
Title: A Multi-center, Phase II Study to Evaluate Efficacy and Safety of Perioperative Chemotherapy With Fluorouracil, Leucovorin, Oxaliplatin, Docetaxel (FLOT) and Trastuzumab in Combination With Toripalimab in Patients With HER2 Positive Locally Advanced Gastric or Esophagogastric Junction Adenocarcinoma
Brief Title: Perioperative Chemotherapy Plus Trastuzumab Plus Toripalimab in HER2 Positive Locally Advanced Gastric or Esophagogastric Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yu jiren (Other)
Responsible Party: Sponsor-Investigator, Yu jiren, Director of gastrointestinal surgery department, First Affiliated Hospital of Zhejiang University
Organization: First Affiliated Hospital of Zhejiang University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20220076C-R1
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Adenocarcinoma of the Stomach; Adenocarcinoma of Esophagogastric Junction; HER2-positive Gastric Cancer
Keywords: Gastric Adenocarcinoma; Esophagogastric Junction Adenocarcinoma; Perioperative Chemotherapy; Trastuzumab; Toripalimab
MeSH Terms: interventions — toripalimab; Trastuzumab; Fluorouracil; Leucovorin; Docetaxel; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: Drug: 5-FU, leucovorin, docetaxel, oxaliplatin (FLOT) Drug: Trastuzumab Drug: Toripalimab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab plus Trastuzumab with FLOT(5-FU+leucovorin+docetaxel+oxaliplatin) (Experimental)
  Interventions: Drug: Toripalimab; Drug: Trastuzumab; Drug: 5-FU, leucovorin, docetaxel, oxaliplatin (FLOT)

INTERVENTIONS:
Drug: Toripalimab — Toripalimab, 240 mg IV infusion on Day 1 of each 21 day cycle for 3 cycles prior to surgery and 3 cycles after surgery.
Drug: Trastuzumab — Trastuzumab, 8 mg/kg IV loading dose at 1st administration and then 6 mg/kg IV on Day 1 of each 21 day cycle for 3 cycles before surgery and 3 cycles after surgery. The first administration of trastuzumab after surgery should also be given at the loading dose of 8 mg/kg.
Drug: 5-FU, leucovorin, docetaxel, oxaliplatin (FLOT) — Pre-operative treatment 4 cycles and post-operative treatment 4 cycles:
  Docetaxel 50 mg/m², IV on day 1 of each 14 day cycle; Oxaliplatin 85 mg/m² , IV on day 1 of each 14 day cycle; Leucovorin 200 mg/m² or Levoleucovorin 100 mg/m², IV on day 1 of each 14 day cycle; 5-FU 2600 mg/m², IV over 24 h on day 1 of each 14 day cycle.

SUMMARY:
This study is a prospective, single arm, multi-center phase II clinical trial designed to evaluate the efficacy and safety of perioperative chemotherapy with FLOT regimen and trastuzumab in combination with toripalimab in participants with resectable HER2 positive locally advanced gastric or esophagogastric junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the clinical study; fully understands and is informed of the study and has signed the Informed Consent Form (ICF).
* The gender is not limited. Age: ≥ 18 years and ≤ 80 years old.
* Gastric or esophagogastric junction adenocarcinoma confirmed by pathology.
* HER2-positive status defined as either IHC score of 3+ or IHC 2+ with amplification proven by fluorescent in situ hybridization (FISH) based on pretreatment endoscopic biopsies.
* Clinical stage at presentation: cT2-T4b, N+/-, M0 as determined by AJCC staging system, 8th edition.

  * The definition of metastatic lymph nodes: a lymph node must be ≥ 10mm in short axis when assessed by CT scan (CT scan slice thickness recommended to be no greater than 5 mm) according to the guideline of Response Evaluation Criteria in Solid Tumours (RECIST version 1.1)
* Participants with a performance status of 0 ~ 1 on the Eastern Cooperative Oncology Group (ECOG) within 7 days before the first dose of study treatment.
* Life expectancy ≥ 6 months.
* Agreement of providing pretreatment endoscopic biopsies specimens and surgical specimens for biomarker analysis, as well as the peripheral blood, feces and urine sample.
* The functions of the vital organs meet requirements as follow (within 14 days before the first dose of study treatment, participant has not received treatment of recombinant human thrombopoietin or granulocyte stimulating factor):

  1. Hematological function：

     * White blood cell count (WBC): 3.5 × 10 ^ 9 / L ~12.0 × 10 ^ 9 / L；
     * Absolute neutrophil count (ANC) ≥ 1.5 × 10 ^ 9 / L；
     * Platelet count (PLT) ≥ 100 × 10 ^ 9 / L；
     * Hemoglobin (Hb) ≥ 90 g / L.
  2. Hepatic function：

     * Total bilirubin (TBIL) ≤ 1.5 × ULN (upper limit of normal);
     * Aspartate aminotransferase (AST) ≤ 2.5 × ULN;
     * Alanine aminotransferase (ALT) ≤ 2.5 × ULN;
     * Albumin (ALB) ≥ 30 g / L.
  3. Renal function：

     * Creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance ≥ 60 ml / min for those with creatinine level > 1.5 × ULN.
  4. Coagulation function：

     * International normalized ratio (INR) ≤ 1.5;
     * Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN.
  5. Cardiac function:

     * The left ventricular ejection fraction (LVEF) value ≥ 55 %, as assessed by echocardiography
* Female of childbearing age must meet requirements: urine or serum pregnancy test must be negative within 7 days before the first dose of study treatment, and she must agree to use adequate contraception methods or keep abstinence (starting with the ICF is signed through 120 days after the last dose of toriplimab, or 210 days after the last dose of trastuzumab, or 180 days after the last dose of chemotherapy, whichever is longer, and should not be breastfeeding. For the male participants must meet requirements: agree to use adequate contraception methods or keep abstinence (starting with the ICF is signed through 120 days after the last dose of toriplimab, or 210 days after the last dose of trastuzumab, or 180 days after the last dose of chemotherapy, whichever is longer).

Exclusion Criteria:

* Prior systemic therapy for treatment of gastric cancer (surgery, chemotherapy, radiotherapy, targeted therapy or immunotherapy).
* Previous or concurrent have other active malignant tumors within the past 5 years (except for basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate cancer or cervical cancer or breast cancer in situ that has undergone curative therapy).
* Participants with gastric outlet obstruction, or unable for oral take, or severe gastrointestinal bleeding.
* Myocardial infarction within 6 months before the first dose of study treatment, uncontrolled angina, arrhythmia which need medical intervention (including but not limited to cardiac pacemaker), congestive heart failure (New York Heart Association (NYHA) class III or IV).
* Existence of chronic diarrhea (watery diarrhea: ≥ 5 times per day).
* Participants with active infection within 14 days before the first dose of study treatment which need medical intervention.
* Participants with active tuberculosis.
* Previous or concurrent diagnosed with interstitial lung disease by imaging or symptoms.
* Any of the following test is positive: Human Immunodeficiency Virus (HIV) antibody, Hepatitis B surface Antigen (HBsAg), or Hepatitis C Virus (HCV) antibody.
* Participants who need long-term systemic steroid therapy (> 10 mg/d prednisone equivalent) or any other form of immunosuppressive therapy within 14 days before the first dose of study treatment or during the study period.
* Concurrent or previous have severe allergic reaction to any antibody-based drugs.
* Existence of any concurrent autoimmune disease, excepting participants with diabetes mellitus type I, hypothyroidism requiring only hormone replacement therapy.
* Receive live vaccines within 28 days before the first dose of study treatment or during the study period, excepting inactivated viral vaccines for seasonal influenza.
* Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* Existence of systemic disease that is difficult to control despite treatment with several agents, for example, diabetes mellitus, hypertension, etc.
* Existence of other serious physical or mental diseases or serious laboratory abnormalities that may increase the risk of participating in the study. Participants who were judged unsuitable as subjects of this trial by investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Rate of pathological complete responses (pCR) | From enrollment to surgery after pre-operative treatment (up to approximately 24 months)
  Percentage of patients with pCR referring to the total number of enrolled and eligible patients, as evaluated centrally by a reference pathologist.

SECONDARY OUTCOMES:
Overall survival | From enrollment to the end of follow up or death from any cause (up to approximately 60 months)
  The duration of overall survival (OS) will be determined by measuring the time interval from enrollment to the end of follow up or death from any cause
Progression-free survival | From enrollment to the end of follow up or the time of disease progression or relapse or death from any cause (up to approximately 60 months)
  Progression-free survival (PFS) will be defined as the time from enrollment to the end of follow up or the time of disease progression or relapse or death from any cause
The incidences and types of adverse events (AE) and severe adverse events (SAE) | From enrollment to 90-day after the last dose administration (up to approximately 27 months)
  The incidences and types of adverse events that occur during treatment will be evaluated according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.3

CONTACTS AND LOCATIONS:
Overall Officials: Jiren Yu, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (8):
- China (8):
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Huzhou Central Hospital, Huzhou, Zhejiang
  - Lishui Central Hospital, Lishui, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Ningbo Medical Center LiHuiLi Hospital, Ningbo, Zhejiang
  - Ningbo Second Hospital, Ningbo, Zhejiang
  - Taizhou Hospital, Taizhou, Zhejiang